CLINICAL TRIAL: NCT01132209
Title: Suture Techniques to Reduce the Incidence of The inCisional Hernia
Acronym: STITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Sint Franciscus Gasthuis (Other); Vlietland Ziekenhuis (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Meander Medical Center (Other); Kennemer Gasthuis (Other); Rijnstate Hospital (Other); Groene Hart Ziekenhuis (Other); Havenziekenhuis (Other); Red Cross Hospital Beverwijk (Other)
Responsible Party: Principal Investigator, joris harlaar, Prof dr JF Lange, professor of Surgery, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STITCH trial MEC 2009-026
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Hernia; Wound Infection; Burst Abdomen; Pain; Quality of Life
Keywords: surgery; incisional hernia; woundinfection; burst abdomen; pain
MeSH Terms: conditions — Hernia; Wound Infection; Pain; Incisional Hernia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Large tissue bites (Active Comparator): As control the conventional large bites technique (mass closure) will be applied in with bites widths of 1 cm and inter-suture spacing of 1 cm with the use of PDS plus ll 1-0 double loop suture material with a 48 mm needle.
  Interventions: Procedure: Closure of the abdominal wall after midline incisions
- small tissue bites (Experimental): In the other group of 288 patients the small bites technique will be applied with bite widths of 0,5 cm and inter suture spacing of 0,5 cm with the use of PDS plus ll 2-0 single suture material with a 31 mm needle placed in the linea alba. In the small bites technique, twice as many stitches will be placed per sutured cm, with a smaller needle and thinner suture material.
  Interventions: Procedure: Closure of the abdominal wall after midline incisions

INTERVENTIONS:
Procedure: Closure of the abdominal wall after midline incisions — Closure of the midline incision after any abdominal operation. Suturing of the fascia of the abdominal wall with two different techniques

SUMMARY:
The objective of the study is reduction of the incidence of the most frequent complication of abdominal surgery, incisional hernia. In this multi center double-blinded prospective randomized controlled trial, in which a new suture technique using small bites is compared with the traditionally applied large bites (mass closure) technique for midline incisions.

ELIGIBILITY:
Inclusion criteria

* Signed informed consent
* All laparotomies with a midline incision
* Age > 18 years

Exclusion criteria

* Previous incisional hernia after midline incision
* Previous surgery through a midline incision within 3 months
* Pregnancy (in women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Incisional hernia occurrence within one year after operation clinical and/or radiographically detected | one year

SECONDARY OUTCOMES:
postoperative complications; in particular wound infection (during admission), burst abdomen (during admission) and wound pain (measured with a visual analog scale (VAS) during the first 6 days after surgery). | one month

CONTACTS AND LOCATIONS:
Overall Officials: Johan Lange, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] Millbourn D, Cengiz Y, Israelsson LA. Effect of stitch length on wound complications after closure of midline incisions: a randomized controlled trial. Arch Surg. 2009 Nov;144(11):1056-9. doi: 10.1001/archsurg.2009.189. PMID 19917943
- [Background] Harlaar JJ, van Ramshorst GH, Nieuwenhuizen J, Ten Brinke JG, Hop WC, Kleinrensink GJ, Jeekel H, Lange JF. Small stitches with small suture distances increase laparotomy closure strength. Am J Surg. 2009 Sep;198(3):392-5. doi: 10.1016/j.amjsurg.2008.10.018. Epub 2009 Mar 12. PMID 19285296
- [Background] Millbourn D, Israelsson LA. Wound complications and stitch length. Hernia. 2004 Feb;8(1):39-41. doi: 10.1007/s10029-003-0159-4. Epub 2003 Sep 6. PMID 13680306
- [Derived] Deerenberg EB, Harlaar JJ, Steyerberg EW, Lont HE, van Doorn HC, Heisterkamp J, Wijnhoven BP, Schouten WR, Cense HA, Stockmann HB, Berends FJ, Dijkhuizen FPH, Dwarkasing RS, Jairam AP, van Ramshorst GH, Kleinrensink GJ, Jeekel J, Lange JF. Small bites versus large bites for closure of abdominal midline incisions (STITCH): a double-blind, multicentre, randomised controlled trial. Lancet. 2015 Sep 26;386(10000):1254-1260. doi: 10.1016/S0140-6736(15)60459-7. Epub 2015 Jul 15. PMID 26188742
- [Derived] Harlaar JJ, Deerenberg EB, van Ramshorst GH, Lont HE, van der Borst EC, Schouten WR, Heisterkamp J, van Doorn HC, Cense HA, Berends F, Stockmann HB, Vrijland WW, Consten EC, Ottow RT, Go PM, Hermans JJ, Steyerberg EW, Lange JF. A multicenter randomized controlled trial evaluating the effect of small stitches on the incidence of incisional hernia in midline incisions. BMC Surg. 2011 Aug 26;11:20. doi: 10.1186/1471-2482-11-20. PMID 21871072